CLINICAL TRIAL: NCT02106208
Title: Study of the Impact of Dairy Fat on Cardiovascular Health.
Acronym: HDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government); Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Benoit Lamarche, PhD, Laval University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: INAF-2013-251
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cheese diet (Experimental): A 4-week experimental diet with all meals and foods be provided to participants, including 90g of regular cheddar cheese daily per 2500 kcal. The diet will contain 13% of saturated fat (SFA), 14% of mono-unsaturated fat (MUFA), 5% of polyunsaturated fat (PUFA) and 53% of carbohydrate (CHO).
  Interventions: Other: Cheese diet
- Butter diet (Experimental): A 4-week experimental diet with all meals and foods be provided to participants, the diet will contain 13% of SFA mostly from butter. The diet will contain 14% of MUFA, 5% of PUFA and 53% of CHO.
  Interventions: Other: Butter diet
- CHO diet (Experimental): A 4-week experimental diet with all meals and foods will provided to participants. The diet will contain 60% of CHO, 6% of SFA, 14% of MUFA and 5% of PUFA.
  Interventions: Other: CHO diet
- MUFA diet (Experimental): A 4-week experimental diet with all meals and foods be provided to participants. The diet will contain 21% of MUFA, 6% of SFA, 5% of PUFA and 53% of CHO.
  Interventions: Other: MUFA diet
- PUFA diet (Experimental): A 4-week experimental diet with all meals and foods will be provided to participants. The diet will contain 12% of PUFA, 14% of MUFA, 6% of SFA and 53% of CHO.
  Interventions: Other: PUFA diet

INTERVENTIONS:
Other: Cheese diet
  Arms: Cheese diet
Other: Butter diet
  Arms: Butter diet
Other: CHO diet
  Arms: CHO diet
Other: MUFA diet
  Arms: MUFA diet
Other: PUFA diet
  Arms: PUFA diet

SUMMARY:
Market trends depicted by Agriculture and Agri-Food Canada suggest stagnation in cheese consumption, with potentially important impact on this key industry in Canada. This is in part due to the commonly accepted notion that saturated fat in the diet, of which cheese contributes significantly, increases the risk of heart disease. Yet, a rather large body of recent evidence suggests that saturated fat may have been unfairly demonized and that its impact on the risk of heart disease may in fact be less important than originally thought. This concept that dairy fat increases the risk of heart attacks therefore needs to be revisited, and this is one of the key objectives of this proposed research program.

The proposed research is designed to investigate for the first time if dairy fat improves the levels of the so-called "good cholesterol", a protective risk factor that has been essentially ignored in the arguments supporting the reduction of saturated fat for heart health.

Our hypothesis is that consumption of SFA from dairy (cheese) compared with a low fat diet and diets rich in MUFA and PUFA leads to favorable changes in plasma HDL-C concentrations and functional characteristics. Consumption of SFA from dairy (cheese) also increases LDL particle size, reduces inflammation and has no deleterious impact on plasma LDL-C and apolipoproteins B (apoB) concentrations compared with a low fat diet.

DETAILED DESCRIPTION:
This is a multi-center randomized crossover controlled feeding study. Briefly, adult men and women will be recruited in the Quebec City and Winnipeg metropolitan area through the media (newspaper, radio), local lipid clinics and mailing lists (n=90).

Participants will be randomized to a series of 5 experimental diets of 4 weeks each: 1- Cheese diet, 2- Butter diet, 3- Carbohydrate (CHO) diet, 4- MUFA diet, 5- PUFA diet. Usual energy intake will be estimated at the beginning of the study using validated tools. Experimental diets will be provided as part of a full feeding protocol under carefully controlled isocaloric conditions to maintain body weight constant. All meals and foods will be provided to participants so that control for energy and macronutrient intake will be optimized. The breakfast meal will represent approximately 30% of the daily energy intake whereas the lunch and dinner meals each will provide 35% of daily energy intake. Participants will be instructed to consume their entire meals. A seven-day cyclic menu will be used. The diets will be separated by washout periods of 4 weeks. Blood samples will be collected on two consecutive days before and after each dietary phase. The mean of the two consecutive measurements will be used in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age between 18 and 65 years
* Waist circumference >80.0 cm for women and >94.0 cm for men
* Plasma concentration of triglycerides >1.70 mmol / L
* Stable weight for 6 months before the start of the study (+/- 5lbs)

Exclusion Criteria:

* Men or women aged under 18 years or over 65 years
* History of CVD, type 2 diabetes or dyslipidaemia monogenic
* Endocrine disorders
* Smoking
* Lipid lowering medications or hypertension medications
* Food allergies and aversions to any food in the composition of experimental menus
* Subjects with special dietary habits (e.g. vegetarianism)
* Subject with a calculated Framingham risk of cardiovascular disease (CVD) > 20%

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in High-Density-Lipoproteins concentrations (HDL-C) | 4 weeks (end-point value)
  Post-diet values will be compared; the primary analysis (pre-determined comparisons) are
  1. Cheese vs Butter,
  2. Cheese vs CHO, MUFA, PUFA
  3. Butter vs. CHO, MUFA, PUFA

SECONDARY OUTCOMES:
Change in HDL-C particle size and subclass | 4 weeks (end-point value)
  Post-diet values will be compared; the primary analysis (pre-determined comparisons) are
  1. Cheese vs Butter,
  2. Cheese vs CHO, MUFA, PUFA
  3. Butter vs. CHO, MUFA, PUFA
Change in HDL cholesterol efflux | 4 weeks (end-point value)
  In a subset of individual;
  Post-diet values will be compared; the primary analysis (pre-determined comparisons) are
  1. Cheese vs Butter,
  2. Cheese vs CHO, MUFA, PUFA
  3. Butter vs. CHO, MUFA, PUFA
Change in Low Density Lipoproteins (LDL) particle size | 4 weeks (end-point value)
  Post-diet values will be compared; the primary analysis (pre-determined comparisons) are
  1. Cheese vs Butter,
  2. Cheese vs CHO, MUFA, PUFA
  3. Butter vs. CHO, MUFA, PUFA
Change in C-Reactive Proteins (CRP) concentrations | 4 weeks (end-point value)
  Post-diet values will be compared; the primary analysis (pre-determined comparisons) are
  1. Cheese vs Butter,
  2. Cheese vs CHO, MUFA, PUFA
  3. Butter vs. CHO, MUFA, PUFA
Change in adiponectin concentrations | 4 weeks (end-point value)
  Post-diet values will be compared; the primary analysis (pre-determined comparisons) are
  1. Cheese vs Butter,
  2. Cheese vs CHO, MUFA, PUFA
  3. Butter vs. CHO, MUFA, PUFA

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (2):
- Canada (2):
  - Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba
  - Institute of Nutrition and Funtional Foods, Québec

REFERENCES:
- [Derived] Brassard D, Arsenault BJ, Boyer M, Bernic D, Tessier-Grenier M, Talbot D, Tremblay A, Levy E, Asztalos B, Jones PJH, Couture P, Lamarche B. Saturated Fats from Butter but Not from Cheese Increase HDL-Mediated Cholesterol Efflux Capacity from J774 Macrophages in Men and Women with Abdominal Obesity. J Nutr. 2018 Apr 1;148(4):573-580. doi: 10.1093/jn/nxy014. PMID 29659963
- [Derived] Brassard D, Tessier-Grenier M, Allaire J, Rajendiran E, She Y, Ramprasath V, Gigleux I, Talbot D, Levy E, Tremblay A, Jones PJ, Couture P, Lamarche B. Comparison of the impact of SFAs from cheese and butter on cardiometabolic risk factors: a randomized controlled trial. Am J Clin Nutr. 2017 Apr;105(4):800-809. doi: 10.3945/ajcn.116.150300. Epub 2017 Mar 1. PMID 28251937